CLINICAL TRIAL: NCT04358068
Title: A Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy of Hydroxychloroquine and Azithromycin to Prevent Hospitalization or Death in Persons With COVID-19
Brief Title: Evaluating the Efficacy of Hydroxychloroquine and Azithromycin to Prevent Hospitalization or Death in Persons With COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment and lack of community enthusiasm
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5395; 38720 (Other: DAIDS-ES Registry Number)
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; SARS-CoV 2
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) (Experimental): Hydroxychloroquine 400 mg (administered as two 200 mg capsules) orally twice daily for 2 doses starting on Day 0, followed by 200 mg (administered as one 200 mg capsule) orally twice daily for 12 doses (6 days), PLUS:
  Azithromycin 500 mg (administered as two 250 mg capsules) orally as a single dose on Day 0, followed by 250 mg (administered as one 250 mg capsule) orally once daily for 4 doses (4 days).
  Interventions: Drug: Hydroxychloroquine (HCQ); Drug: Azithromycin (Azithro)
- Arm B: Placebo for Hydroxychloroquine and Azithromycin (Placebo Comparator): Placebo for Hydroxychloroquine (administered as two matching placebo capsules) orally twice daily for 2 doses starting on Day 0, followed by Placebo for HCQ (administered as one 200 mg capsule) orally twice daily for 12 doses (6 days), PLUS:
  Placebo for Azithromycin (administered as two matching placebo capsules) orally as a single dose on Day 0, followed by Placebo for Azithromycin (administered as one matching placebo capsule) orally once daily for 4 doses (4 days).
  Interventions: Drug: Placebo for Hydroxychloroquine; Drug: Placebo for Azithromycin

INTERVENTIONS:
Drug: Hydroxychloroquine (HCQ) — Administered orally
  Arms: Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro)
Drug: Azithromycin (Azithro) — Administered orally
  Arms: Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro)
Drug: Placebo for Hydroxychloroquine — Administered orally
  Arms: Arm B: Placebo for Hydroxychloroquine and Azithromycin
Drug: Placebo for Azithromycin — Administered orally
  Arms: Arm B: Placebo for Hydroxychloroquine and Azithromycin

SUMMARY:
The purpose of this study was to evaluate the efficacy of hydroxychloroquine (HCQ) and azithromycin (Azithro) to prevent hospitalization or death in symptomatic adult outpatients with COVID-19 caused by SARS-CoV-2 infection.

DETAILED DESCRIPTION:
This Phase IIB study was designed to evaluate the efficacy of hydroxychloroquine (HCQ) and azithromycin (Azithro) to prevent hospitalization or death in symptomatic adult outpatients with COVID-19 caused by SARS-CoV-2 infection.

Participants were randomized 1:1 to receive active or placebo study treatment. The target sample size was 2000 participants, with approximately 1000 in each arm. Stratification was by "high" versus "low" risk of progression to severe COVID-19, where "high risk" was defined as a person age ≥60 years or having at least one of several specified comorbidities.

Participants were prescribed study treatment for 7 days and were to be followed for an additional 24 weeks. Assessments on a subset of participants were planned to include blood collection, self-collected nasal swabs, and nasopharyngeal swabs.

On June 23, 2020, sites were informed that the study was closing to follow-up due to slow enrollment and lack of community enthusiasm. Follow-up through week 24 was not completed for any participant. Participants were asked to complete the Day 20 visit and then were discontinued from the study. Due to the early termination, enrollment into the specimen collection subset did not occur, and results associated with those specimens are not available. Due to the small number of participants enrolled, some statistical tests were not able to be performed and only descriptive results are provided.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of confirmed active severe acute respiratory syndrome coronavirus (SARS-CoV-2) infection from any respiratory specimen collected ≤7 days from when the first dose of study treatment was expected to be taken.
* Experienced at least one of the following SARS-CoV-2 infection symptoms within 24 hours of screening (symptom(s) must be new or worse compared to pre-COVID-19 health status):

  * Fever (can be subjective) or feeling feverish
  * Cough
  * Shortness of breath or difficulty breathing at rest or with exertion
  * Sore throat
  * Body pain or muscle pain
  * Fatigue
  * Headache
* Agreed to not participate in another clinical trial for the treatment of COVID-19 or SARS-CoV-2 during the study period up until reaching hospitalization or 20 days, whichever is earliest.
* Agreed to not obtain study medications outside of the A5395 study.

Exclusion Criteria:

* Need for hospitalization or immediate medical attention in the clinical opinion of the study investigator.
* History of or current hospitalization for COVID-19.
* History of ventricular arrhythmia or use of antiarrhythmics within 30 days prior to entry.
* Personal or family history of Long QT syndrome.
* History of kidney disease.
* History of ischemic or structural heart disease.
* History of hypokalemia or hypomagnesemia or taking potassium supplementation or magnesium supplementation
* Personal medical history of porphyria, retinopathy, severe hepatic impairment, or glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Used drugs with possible anti-SARS-CoV-2 activity within 30 days prior to study entry, e.g., remdesivir, lopinavir/ritonavir fixed dose combination, ribavirin, chloroquine, hydroxychloroquine, and azithromycin, or participation in a clinical trial involving any of these drugs whether for treatment or prophylaxis.
* Requirement or expected requirement for a medication that significantly prolongs QT intervals or increases risk for QT prolongation.
* Loop diuretics are exceptions to above exclusion criterion but these cannot be used within 30 days prior to study entry.
* Participated in a study where co-enrollment was not allowed.
* Receipt of a SARS-CoV-2 vaccination prior to study entry.
* Known allergy/sensitivity or any hypersensitivity to components of HCQ, azithromycin, or their formulation.
* More than 10 days of any of the following symptoms attributed to the SARS-CoV-2 infection at study entry:

  * Fever (can be subjective) or feeling feverish
  * Cough
  * Shortness of breath or difficulty breathing at rest or with exertion
  * Sore throat
  * Body pain or muscle pain
  * Fatigue
  * Headache
  * Chills
  * Nasal obstruction or congestion
  * Loss of taste or smell
  * Nausea or vomiting
  * Diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davey Smith, MD, Study Chair — University of California, San Diego
Locations (11):
- United States (11):
  - Alabama CRS, Birmingham, Alabama
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Harbor-UCLA CRS, Torrance, California
  - Whitman-Walker Health CRS, Washington D.C., District of Columbia
  - Northwestern University CRS, Chicago, Illinois
  - Rush University CRS, Chicago, Illinois
  - Greensboro CRS, Greensboro, North Carolina
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - Trinity Health and Wellness Center CRS, Dallas, Texas
  - University of Washington AIDS CRS, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://submit.mis.s-3.net/ Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.

REFERENCES:
- See also: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (Corrected Version 2.1 - July 2017) — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between 13MAY2020 and 15JUN2020 at US based clinical research sites
Groups:
- Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro): Hydroxychloroquine 400 mg (administered as two 200 mg capsules) orally twice daily for 2 doses starting on Day 0, followed by 200 mg (administered as one 200 mg capsule) orally twice daily for 12 doses (6 days), PLUS:
  Azithromycin 500 mg (administered as two 250 mg capsules) orally as a single dose on Day 0, followed by 250 mg (administered as one 250 mg capsule) orally once daily for 4 doses (4 days).
  Hydroxychloroquine (HCQ): Administered orally
  Azithromycin (Azithro): Administered orally
- Arm B: Placebo for Hydroxychloroquine and Azithromycin: Placebo for Hydroxychloroquine (administered as two matching placebo capsules) orally twice daily for 2 doses starting on Day 0, followed by Placebo for HCQ (administered as one 200 mg capsule) orally twice daily for 12 doses (6 days), PLUS:
  Placebo for Azithromycin (administered as two matching placebo capsules) orally as a single dose on Day 0, followed by Placebo for Azithromycin (administered as one matching placebo capsule) orally once daily for 4 doses (4 days).
  Placebo for Hydroxychloroquine: Administered orally
  Placebo for Azithromycin: Administered orally
Period: Overall Study
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin
Started (Indicates the number randomized to a given arm) | 9 | 11
Completed | 7 | 9
Not Completed | 2 | 2
Not completed — Did not initiate study treatment | 2 | 2

BASELINE CHARACTERISTICS:
Population: Participants who initiated study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Median (Full Range); unit: years] | 44 [30 to 61] | 35 [30 to 49] | 39 [30 to 61]
Age, Customized [Count of Participants; unit: Participants]
  < 60 years | 5 | 9 | 14
  >= 60 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 0 | 5 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 9 | 16
Risk of progression to severe disease [Count of Participants; unit: Participants] — "High" risk is defined by any of the following: Aged 60 years and older; Chronic lung disease or moderate to severe asthma; Immunocompromised status due to disease (ex. those living with HIV with a CD4+ T-cell count of <200/mm^3); Immunocompromised status due to medication (ex. persons taking 20 mg or more of prednisone equivalents a day, anti-inflammatory monoclonal antibody therapies, or cancer therapies); Severe obesity (body mass index [BMI] >40 kg/m^2); Hypertension; Cardiovascular disease; Diabetes; Chronic kidney disease; Chronic liver disease
  Participants
    High risk | 4 | 2 | 6
    Low risk | 3 | 7 | 10
Time from symptom onset to treatment start [Median (Full Range); unit: days] | 5 [4 to 8] | 4 [3 to 20] | 5 [3 to 20]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Died From Any Cause or Were Hospitalized
Description: Hospitalization was defined as requiring at least 24 hours of acute care in a hospital or similar acute care facility, including Emergency Rooms or temporary facilities instituted to address needs during the COVID-19 pandemic. Evaluation at a hospital or similar facility with less than 24 hours of acute care was not considered a hospitalization. Formal statistical testing was not conducted due to the small number of participants and events.
Time Frame: The 20-day period from and including the day of the first dose of study treatment
Population: Participants who initiated study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin
Number analyzed (Participants) | 7 | 9
Participants | 0 | 1

2. Secondary Outcome: Number of Participants Who Died From Any Cause
Description: Deaths reported due to any cause (COVID-related or not)
Time Frame: The 20-day period from and including the day of the first dose of study treatment
Population: Participants who initiated study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin
Number analyzed (Participants) | 7 | 9
Participants | 0 | 0

3. Secondary Outcome: Number of Participants Who Died From Any Cause, or Were Hospitalized, or Had an Urgent Visit to Emergency Room or Clinic
Description: Hospitalization was defined as requiring at least 24 hours of acute care in a hospital or similar acute care facility, including Emergency Rooms or temporary facilities instituted to address needs during the COVID-19 pandemic. Evaluation at a hospital or similar facility with less than 24 hours of acute care was not considered a hospitalization, but was included for this outcome measure.
Time Frame: The 20-day period from and including the day of the first dose of study treatment
Population: Participants who initiated study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin
Number analyzed (Participants) | 7 | 9
Participants | 1 | 1

4. Secondary Outcome: Number of Participants Who Died From Any Cause or Were Hospitalized Through the End of Follow-up
Description: Hospitalization was defined as requiring at least 24 hours of acute care in a hospital or similar acute care facility, including Emergency Rooms or temporary facilities instituted to address needs during the COVID-19 pandemic. Evaluation at a hospital or similar facility with less than 24 hours of acute care was not considered a hospitalization. Due to the early termination of the study, participant followup was discontinued at Day 20. Refer to the primary outcome above for results based on the time frame out to Day 20.
Time Frame: From day of the first dose of study treatment to Week 24
Population: Due to the early termination of the study, the data were not collected
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants Who Prematurely Discontinue Study Treatment Due to an Adverse Event
Description: Premature discontinuation of study treatment is defined as a permanent discontinuation of either study treatment (HCQ/Placebo and/or Azithro/Placebo)
Time Frame: From start of study treatment through Day 7
Population: Participants who initiated study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin
Number analyzed (Participants) | 7 | 9
Participants | 0 | 1

6. Secondary Outcome: Number of Participants Who Had Any Cardiac Adverse Events
Description: Cardiac adverse events included in the analysis were chosen a priori by the study chairs
Time Frame: From start of study treatment through Day 20
Population: Participants who initiated study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin
Number analyzed (Participants) | 7 | 9
Participants | 0 | 0

7. Secondary Outcome: Duration of Fever
Description: Defined as the time from study treatment initiation to the last day in the participant's daily diary card on which a temperature greater than 100.4°F was recorded or a potentially antipyretic drug, such as acetaminophen or ibuprofen, was taken. Participants with at least one temperature who never reported fever or use of anti-pyretic medications were assigned a duration of zero days
Time Frame: Day 0 to Day 20, 21 days total
Population: Participants who initiated study treatment and reported at least one temperature on the diary card
Measure: Median (Full Range); unit: days
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin
Number analyzed (Participants) | 7 | 8
days | 0 [0 to 7] | 0 [0 to 4]
Statistical Analysis 1: Comparison: Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) vs Arm B: Placebo for Hydroxychloroquine and Azithromycin; Test type: Superiority — Participant specific durations were compared between randomized arms using a two-sided Wilcoxon test with a two-sided 5% type I error rate; p = 0.51, Wilcoxon (Mann-Whitney) — Wilcoxon Test was not stratified by high/low risk because of the small number enrolled

8. Secondary Outcome: Duration of Symptoms Associated With COVID-19 Disease
Description: Defined as the time from start of study treatment to the last day in the participant's daily diary card on which a moderate or worse targeted symptom was recorded. The set of target symptoms were cough, shortness of breath, feeling feverish, fatigue, muscle aches, diarrhea, vomiting, nausea, headache, sore throat, nasal obstruction (stuffy nose), nasal discharge (runny nose), loss of smell, and loss of taste. Participants who had missing diary records due to hospitalization were assumed to have moderate symptoms during the period of hospitalization in the analysis. Missing diary card records not due to hospitalization were assumed to have absent symptoms.
Time Frame: Day 0 to Day 20, 21 days total
Population: Participants who initiated study treatment
Measure: Median (Full Range); unit: days
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin
Number analyzed (Participants) | 7 | 9
days | 11.0 [5.0 to 17.0] | 10.0 [5.0 to 21.0]
Statistical Analysis 1: Comparison: Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) vs Arm B: Placebo for Hydroxychloroquine and Azithromycin; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.79, Wilcoxon (Mann-Whitney) — Wilcoxon Test was not stratified by high/low risk because of the small number enrolled

9. Secondary Outcome: Participant-specific Area Under the Curve (AUC) of the Symptom Score Associated With COVID-19 Disease Over Time
Description: Defined as the sum of scores for the targeted symptoms (defined in the protocol) in the participant's daily diary record (each symptom was scored from 0-best to 3-worst). Participant-specific areas under the curve (AUC) over time were calculated using the trapezoidal rule and defined as the area below the line formed by joining total symptom scores on each daily diary card from the pre-treatment score on Day 0 through to Day 20. AUCs were rescaled by time by dividing by 21 (corresponding to the number of daily diary cards during follow-up between pre-treatment Day 0 and Day 20), in order to provide results on a symptom scale from 0-best to 42-worst (for non-hospitalized participants). Participants who were hospitalized were assigned a value equal to the sum of the maximum possible scaled AUC (42) and the duration of hospitalization, and thus values >42 were possible. Missing scores between pre-treatment and Day 20 were linearly interpolated. Higher AUCs indicate worse outcomes.
Time Frame: Day 0 to Day 20, 21 days total
Population: Participants who initiated study treatment
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin
Number analyzed (Participants) | 7 | 9
score on a scale | 4.0 [0.9 to 18.0] | 2.8 [0.5 to 46.0]
Statistical Analysis 1: Comparison: Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) vs Arm B: Placebo for Hydroxychloroquine and Azithromycin; Test type: Superiority — Participant specific AUCs were compared between randomized arms using a two-sided Wilcoxon test with a two-sided 5% type I error rate; p = 0.53, Wilcoxon (Mann-Whitney) — Wilcoxon Test was not stratified by high/low risk because of the small number enrolled

10. Secondary Outcome: Time to Self-reported Return to Usual (Pre-COVID) Health.
Description: Time to self-reported return to (pre-COVID) usual health was defined as the time from the start of study treatment to the first day in the participant's daily diary card on which they responded 'Yes' with no subsequent reports of 'No' to the question "Have you returned to your usual (pre-COVID) health today?" Participants who never reported a 'Yes' response were assigned a duration of 22 days.
Time Frame: Day 0 to Day 20, 21 days total
Population: Participants who initiated study treatment
Measure: Median (Full Range); unit: days
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin
Number analyzed (Participants) | 7 | 9
days | 17.0 [6.0 to 22.0] | 10.0 [6.0 to 22.0]
Statistical Analysis 1: Comparison: Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) vs Arm B: Placebo for Hydroxychloroquine and Azithromycin; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.83, Wilcoxon (Mann-Whitney) — Wilcoxon Test was not stratified by high/low risk because of the small number enrolled

11. Secondary Outcome: SARS-CoV-2 RNA Detection Status From Self-collected Nasal and Site-collected NP Swabs Among Subset
Description: The virology substudy did not open to enrollment and thus no data on virologic outcomes are available to report
Time Frame: Measured at entry, Day 6, and Day 20
Population: The virology substudy did not open to enrollment and thus no data on virologic outcomes are available
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: SARS-CoV-2 RNA Level (Continuous) From Self-collected Nasal and Site-collected NP Swabs Among Subset
Description: The virology substudy did not open to enrollment and thus no data on virologic outcomes are available to report
Time Frame: Measured at entry, Day 6, and Day 20
Population: The virology substudy did not open to enrollment and thus no data on virologic outcomes are available to report
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Participants With an Occurrence of Fainting
Description: Fainting was self-reported on the study diary card as absent (score 0), mild (1), moderate (2), or severe (3); scores of > 0 are defined as an occurrence of fainting
Time Frame: From start of study treatment through Day 20
Population: Participants who initiated study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin
Number analyzed (Participants) | 7 | 9
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: From enrollment to the end of follow up (Participants were asked to complete the Day 20 visit and then were discontinued from the study)
Description: Post-entry adverse event (AE) reporting requirements were: All Grade ≥3 AEs; All cardiac AEs regardless of grade; All AEs that led to a change in study treatment/intervention regardless of grade; All AEs meeting SAE definition or EAE reporting requirement. DAIDS AE Grading Table, Version 2.1 and DAIDS EAE Manual Version 2.0 were used for this study.
Arm/Group | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) | Arm B: Placebo for Hydroxychloroquine and Azithromycin
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/11
Other Adverse Events (participants affected / at risk) | 2/9 | 3/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) (N=9) | Arm B: Placebo for Hydroxychloroquine and Azithromycin (N=11)
COVID-19 (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Hydroxychloroquine (HCQ) and Azithromycin (Azithro) (N=9) | Arm B: Placebo for Hydroxychloroquine and Azithromycin (N=11)
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Ageusia (Nervous system disorders) | 1 | 1
Anosmia (Nervous system disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to slow enrollment and lack of community enthusiasm. Follow-up through week 24 was not completed for any participant. Participants were asked to complete the Day 20 visit and then were discontinued from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT04358068/Prot_002.pdf
  • Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT04358068/SAP_001.pdf
  • Informed Consent Form (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT04358068/ICF_000.pdf